CLINICAL TRIAL: NCT01807962
Title: A Randomised Double Blind Controlled Trial of Injection of Local Anaesthetic and Corticosteroid Under Ultrasound Control in the Greater Trochanteric Pain Syndrome.
Brief Title: Local Injection Under US Control in GTPS.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slower than planned recruitement
Sponsor: Stephane Genevay (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Stephane Genevay, Médecin adjoint, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CE 10-213
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Periarthritis; Bursitis
Keywords: Injections, Subcutaneous; Cortisone; Anesthetics, Local
MeSH Terms: conditions — Periarthritis; Bursitis | interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rapidocain and bethametsaone (Active Comparator): Rapidocain and Bethametsaone :
  Lidocaine (Rapidocain(R)): 4ml of 1% Lidocaine Bethametasone (Diprophos): 1ml ampoule (containing 5mg/ml dipropionate de bétaméthasone and 2mg/ml phosphate disodique de bétaméthasone)
  Interventions: Drug: rapidocain and bethametsaone
- sterile saline (Placebo Comparator): Placebo arm with 5ml of sterile saline (NaCl) solution
  Interventions: Drug: sterile saline

INTERVENTIONS:
Drug: rapidocain and bethametsaone — lidocaine (Rapidocain(R)): 4ml of 1% Lidocaine
  bethametasone (Diprophos): 1ml ampoule (containing 5mg/ml dipropionate de betamethasone and 2mg/ml phosphate disodique de betamethasone)
  Other Names: diprophos; lidocaine
  Arms: rapidocain and bethametsaone
Drug: sterile saline — Placebo = 5ml of sterile saline solution
  Other Names: NaCl
  Arms: sterile saline

SUMMARY:
We hypothesize that local ultrasound guided injection with corticosteroid and local anaesthetic are effective on the symptoms of GTPS.

DETAILED DESCRIPTION:
The greater trochanteric pain syndrome (GTPS) is a frequent soft tissue syndrome which is often not recognised by medical practitioners. Currently, there is no validated definition of this syndrome and it is classically defined as pain and tenderness in the region of the greater trochanter that may radiate down to the postero-lateral aspect of the thigh and may mimic nerve root compression.

The prevalence of GTPS amongst adult patients referred to a spine clinic for chronic low back pain (LBP) has been reported to be 20-35%. In addition to pain, GTPS induces functional disability which at times may profoundly interfere with patients' daily activities. The diagnosis of GTPS is suspected in a patient complaining of lateral hip pain. The reproduction of typical pain on palpation of the posterior part of the greater trochanter is the only well recognised clinical sign, although other clinical signs have been described. As is frequently the case with these type of syndromes, the physiopathology of GTPS is probably a mixture of several musculoskeletal problems, among which trochanteric bursitis and gluteus medius (GMe) tendinosis are the most frequently cited.

MRI studies have demonstrated GMe tendinosis or tears in patients with GTPS and MRI is used as the gold standard for the diagnosis of GTPS in many studies. Musculoskeletal ultrasound (US) is of increasing interest among rheumatologists. It readily demonstrates soft tissue lesions, fluid collections, allows dynamic examination and the undertaking of ultrasound guided procedures. GMe and gluteus minus (GMi) tendinopathy or tears as well as bursitis can be clearly demonstrated by ultrasound and US may guide steroid injection for the treatment of GMe tendinopathy. However, to date no study has compared the utility of MRI compared to US.

There are very few well-performed studies regarding the treatment of GTPS. Although poorly studied, analgesics and non steroidal anti-inflammatory drugs (NSAIDs) are often used as first line therapy. The duration of therapy required with these oral agents is unknown and there are significant potential side-effects from these treatments. The vast majority of patients referred to secondary or tertiary centres have failed these oral therapies. Some authors advocate physiotherapy (massage or stretching) but once again, there is no strong evidence to support this approach. Thus, most patients are treated with an injection of a combination of steroids and local anaesthetic. However, there is no convincing evidence in the literature that this practice is effective.

The use of musculoskeletal ultrasound (US) has been shown to improve the accuracy of corticosteroid injections for many joints and extra-articular structures such as bursa and tendon sheaths. Although small observational studies have suggested that local corticosteroid injection may be effective in the short term, no prospective controlled study has been carried out to establish the efficacy of this common intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients complaining of lateral hip pain for more than 1 month.
2. NRS lateral hip pain score ≥ 4 in the preceding week.
3. Failure of another "standard" treatment:

   * Physiotherapy: local therapy or a stretching program, or
   * Analgesic treatment (minimum of 5 days of consecutive therapy, including, but not limited to, NSAIDs).
4. Typical lateral hip pain reproduced by palpation of the greater trochanter

Exclusion Criteria:

1. Age younger than 18 years old
2. Concomitant local surgical intervention for tumours, infection or fracture, based on clinical history and physical examination
3. Previous ipsilateral prosthetic hip surgery
4. Scheduled ipsilateral hip surgery within 3 months
5. Fibromyalgia (diagnosis established by a rheumatologist)
6. Flair of chronic inflammatory joint disease (as defined by a rheumatologist)
7. Skin lesions at the injection site
8. Allergy to one of the studied drugs
9. Anticoagulation with internal normalized ration (INR) >3
10. Blood coagulation disorder, such as haemophilia.
11. Serious and uncontrolled psychiatric disease (as assessed by the clinician as a contraindication for steroid)
12. Other contraindications to steroid use, such as:

    * uncontrolled diabetes (non-fasting blood glucose > 10 mmol/L)
    * unstable hypertension (systolic pressure > 160mmHg or diastolic pressure > 100mmHg), or
    * open or closed angle glaucoma.
13. Requirement for systemic steroids (including steroid injections) or dose modification of disease modifying anti-rheumatic drugs during the preceding three months. Oral corticosteroids (< 10mg / day of Prednisone or equivalent) will be permitted providing that the dose has been stable for 4 weeks prior to inclusion and that the patient is expected to remain on the baseline dose for the duration of the study.
14. Presence of a pacemaker or other metallic object that constitutes a CI to MRI, or severe claustrophobia
15. Pregnant women (according to a pregnancy test) or nursing (breastfeeding) mothers.
16. Unwillingness or inability to give informed consent.
17. Unavailability for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of ultrasound-guided injection with corticosteroid and local anaesthetic for GTPS. | 4 weeks
  Difference in pain intensity in the lateral hip region at 4 weeks between the 2 treatment groups, as measured by a NRS. Because the timing of the response to an infiltration is not well established we plan to examine pain both at 4 weeks, as well as longitudinally over 4 weeks(evolution of pain over time).

SECONDARY OUTCOMES:
Number of "responders" | 4 weeks
  Number of "responders" (defined as a reduction in NRS ≥ 1.5)at 4 weeks and at 6 months.
Number of patients with "low residual disease activity" | 4 weeks
  Number of patients with "low residual disease activity" (defined as NRS
  ≤ 2.0)at 4 weeks and at 6 months.
PGI patient | 4 weeks
  Patient Global Assessment
Lumbar spine function | 4 weeks
  Lumbar spine function measured with the Oswestry questionnaire at 4 weeks and at 6 months
Hip joint function | 4 weeks
  Hip joint function (Womac questionnaire)at 4 weeks and 6 months
QoL | 4 weeks
  Quality of life (SF-12)at 4 weeks and 6 months
Requirement for oral analgesics | 4 weeks
  Recording patient requirements for analgesics at weekly intervals following the intervention
Side effects of the intervention | 4 weeks
  Clinical side effects - patients will be questioned specifically with respect to certain side-effects potentially linked to the injection technique and /or the injected substances. Any other side-effects cited by the patient will be recorded appropriately.
  Ultrasound-measured side-effects: hematoma, GMe or GMi tear, tendinosis or calcification post-intervention that had not been visualised on the initial US prior to the first injection.
  Measured at 4 weeks and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Genevay, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided